CLINICAL TRIAL: NCT02652390
Title: Extended Follow-up of a Randomized Placebo-controlled Trial of Local Steroid Injection in Carpal Tunnel Syndrome
Brief Title: Local Steroid Injection vs Placebo in Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Isam Atroshi, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLM_CTS_2
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Methylprednisolone; Methylprednisolone Acetate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methylprednisolone 80 mg (Experimental): Local injection of 80 mg Methylprednisolone into the carpal tunnel
  Interventions: Drug: Methylprednisolone 80 mg
- Methylprednisolone 40 mg (Experimental): Local injection of 40 mg Methylprednisolone into the carpal tunnel
  Interventions: Drug: Methylprednisolone 40 mg
- Placebo (Placebo Comparator): Local injection of saline into the carpal tunnel
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Methylprednisolone 80 mg — 2 mL methylprednisolone (40 mg/mL) + 1 mL lidocaine
  Other Names: Depo-Medrol
  Arms: Methylprednisolone 80 mg
Drug: Methylprednisolone 40 mg — 1 mL methylprednisolone (40 mg/mL) + 1 mL saline + 1 mL lidocaine
  Other Names: Depo-Medrol
  Arms: Methylprednisolone 40 mg
Other: Saline — 2 mL saline + 1 mL lidocaine
  Other Names: Sodium chloride solution
  Arms: Placebo

SUMMARY:
Between 2008 and 2012 the investigators performed a single-center randomized double-blind placebo-controlled trial to assess the efficacy of local injection of two different doses of methylprednisolone (80 mg and 40 mg) in patients with carpal tunnel syndrome (CTS), aged 18 to 70 years, not previously treated with steroid injection. The primary outcomes were change in the CTS symptom severity score at 10 weeks and rate of carpal tunnel release surgery on the study hand at 1 year. In the trial 111 patients were randomized (37 in each of the 3 groups: 80 mg methylprednisolone, 40 mg methylprednisolone and placebo) and all completed the 1-year follow-up. The investiators plan an extended follow-up 5 to 7 years after injection.

DETAILED DESCRIPTION:
Extended follow-up protocol:

All 111 trial participants will be contacted by telephone by a researcher and given information about this extended follow-up. A questionnaire together with written information and consent forms will be sent by mail. The questionnaire consists of the CTS symptom severity sale, 11-item DASH scale, bodily pain scale, and a treatment satisfaction visual analog scale (VAS), that were used in previous follow-up evaluations. The questionnaire will also include the 6-item CTS symptoms scale (CTS-6) and the palmar pain scale. The patients will be asked whether and when they had undergone carpal tunnel release surgery on the study hand after they received the injection within the trial. Patients' records will be reviewed to verify data about subsequent surgery on the study hand.

The Chi-square test will be used to compare the 80-mg methylprednisolone group and the placebo group with regard to the proportion of patients who have had carpal tunnel release surgery on the study hand within 5 years after injection (primary outcome). The change in symptom severity score in patients in the 80-mg methylprednisolone group who did not have surgery on the study hand after injection will be compared with the change in symptom severity score in patients who had surgery on the study hand after methylprednisolone injection (co-primary outcome) using analysis of covariance (ANCOVA) adjusting for sex, age, dominance of the study hand and baseline symptom severity score. A similar comparison will be made for the 11-item DASH and the bodily pain scores. The palmar pain score at 5 to 7 years will be compared between the groups using the independent-samples t-test and also ANCOVA to adjust for sex, age and dominance of the study hand. Patients who had surgery after methylprednisolone injection will be compared with patients who had surgery after placebo injection with regard to change from baseline to 5 to 7 years in the symptom severity score, 11-item DASH scale score, bodily pain score and satisfaction score using ANCOVA adjusting for sex, age, dominance of the study hand and respective baseline score. To identify potential predictive factors for long-term benefit after 80 mg methylprednisolone injection, surgery within 5 years will be analyzed according to the variables sex, age, dominance of the study hand, baseline symptom severity score (≥3 versus < 3) and baseline median nerve conduction abnormality (severe/moderate vs mild/normal).

All statistical tests will be 2-sided and a p value of less than 0.05 will indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Primary idiopathic CTS
* Symptoms of classic or probable CTS according to the Katz diagnostic criteria (numbness and/or tingling in at least 2 of the 4 median nerve innervated fingers)
* Failed treatment with wrist splinting (2 months)
* Nerve conduction tests showing median neuropathy at the wrist or, if normal, two orthopedic surgeons independently make CTS diagnosis
* Symptom severity that warranted referral for consideration for surgery

Exclusion Criteria:

* Previous steroid injection for CTS
* Thenar muscle atrophy
* Sensory deficit (two-point discrimination >8 mm)
* Diabetes, thyroid disorder, or inflammatory disease
* Polyneuropathy or vibration-induced neuropathy
* Current pregnancy
* Previous carpal tunnel surgery on the study hand
* Surgery on the contralateral hand in the past 2 months
* Inability to respond to questionnaires
* Severe medical illness
* Known drug/alcohol abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

REFERENCES:
- [Result] Atroshi I, Flondell M, Hofer M, Ranstam J. Methylprednisolone injections for the carpal tunnel syndrome: a randomized, placebo-controlled trial. Ann Intern Med. 2013 Sep 3;159(5):309-17. doi: 10.7326/0003-4819-159-5-201309030-00004. PMID 24026316
- [Derived] Hofer M, Ranstam J, Atroshi I. Extended Follow-up of Local Steroid Injection for Carpal Tunnel Syndrome: A Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2130753. doi: 10.1001/jamanetworkopen.2021.30753. PMID 34677593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a long-term follow-up of patients who participated in a randomized trial. In the initial trial the patients were recruited between November 7, 1998 and March 10, 2011 (NCT00806871; see Atroshi et al. Ann Intern Med 2013). Data in this follow-up were collected between February 24, 2016 and July 7, 2016.
Pre-assignment Details: No significant events occurred after participant enrollment but prior to assignment to arms.
Period: Overall Study
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo
Started | 37 | 37 | 37
Completed | 37 | 37 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo | Total
Number analyzed (Participants) | 37 | 37 | 37 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at follow-up
  years | 53 (12) | 50 (11) | 55 (12) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 28 | 81
  Male | 11 | 10 | 9 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 37 | 37 | 37 | 111
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 37 | 37 | 37 | 111
Dominant hand treated [Count of Participants; unit: Participants] | 30 | 29 | 28 | 87
Body mass index [Mean (Standard Deviation); unit: kg/m2] — BMI at follow-up
  kg/m2 | 27.3 (4.2) | 27.6 (4.3) | 27.7 (5.7) | 27.5 (4.8)
Follow-up time from randomization/treatment [Mean (Standard Deviation); unit: months] | 74 (7.5) | 74 (7.1) | 74 (7.1) | 74 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Have Had Carpal Tunnel Release Surgery on the Study Hand
Description: Number of patients who have had carpal tunnel release surgery on the study hand.
Time Frame: 5 to 7 years
Population: Data from all trial participants were available with no withdrawals, drop-outs or missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo
Number analyzed (Participants) | 37 | 37 | 37
Participants | 31 | 34 | 36

2. Primary Outcome: Symptom Severity Score
Description: Change in symptom severity score from baseline to 5 to 7 years. Score range 1 (no symptoms) to 5 (most severe symptoms).
Time Frame: 5-7 years
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 80-mg Mrthylprednisolone and no Surgery: Patients in the 80-mg methylprednisolone group who had not undergone carpal tunnel release surgery on the study hand
- Surgery After Methylprednisolone or Placebo: Patients in the methylprednisolone or placebo groups who had undergone carpal tunnel release surgery after injection.
Arm/Group | 80-mg Mrthylprednisolone and no Surgery | Surgery After Methylprednisolone or Placebo
Number analyzed (Participants) | 6 | 101
score on a scale | 1.34 (0.9) | 1.53 (0.9)

3. Secondary Outcome: Palmar Pain Score
Description: Score for pain in the proximal palm and related activity limitations, range 0 (worst) to 100 (best).
Time Frame: 5-7 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo
Number analyzed (Participants) | 37 | 37 | 37
score on a scale | 86.4 (18) | 84.6 (22) | 83.0 (25)

4. Secondary Outcome: 11-item Disabilities of the Arm, Shoulder and Hand (DASH) Score
Description: Score for the 11-item DASH scale, a measure of activity limitations related to the upper extremity. Score range 0 (best) to 100 (worst)
Time Frame: 5-7 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo
Number analyzed (Participants) | 37 | 37 | 37
score on a scale | 13.1 (18) | 16.9 (20) | 19.3 (20)

5. Secondary Outcome: Bodily Pain Score
Description: Score for the 2-item bodily pain scale, range 0 (worst) to 100 (best).
Time Frame: 5-7 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo
Number analyzed (Participants) | 37 | 37 | 37
score on a scale | 81.4 (24) | 79.9 (24) | 78.2 (25)

6. Secondary Outcome: Satisfaction Score
Description: Visual analog scale about treatment satisfaction, score 0 (worst) to 100 (best).
Time Frame: 5-7 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo
Number analyzed (Participants) | 37 | 37 | 37
score on a scale | 77.5 (28) | 71.4 (27) | 68.4 (28)

ADVERSE EVENTS:
Time Frame: 5 to 7 years
Description: Adverse events from patient-reporting and review of medical records.
Arm/Group | Methylprednisolone 80 mg | Methylprednisolone 40 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes